CLINICAL TRIAL: NCT05468125
Title: Special Maternal Care Bundle to Attenuate Spinal Induced Hypotension in Cesarean Section
Brief Title: Maternal Care Bundle to Attenuate Hypotension in Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, Abdelrhman Alshawadfy, Lecturer of anesthesia and intensive care, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Maternal care bundle
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Hypotension; Cesarean Section Complications
MeSH Terms: conditions — Hypotension | interventions — Counseling

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: patients will be randomly allocated by a computer software program (www. Randmizer.org) and allocation sequence will be done by opaque closed envelope.
  Data will be collected by a separate anesthesiologist not sharing in the study and blinded to the technique being used.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- care bundle (Active Comparator): will be subjected to a bundle of care of four elements
  Interventions: Procedure: guidance
- best-evidenced practice (Active Comparator): will be guided according to the best-evidenced performance consisting of three elements
  Interventions: Procedure: guidance

INTERVENTIONS:
Procedure: guidance — either follow the care bundle or the best evidence practice

SUMMARY:
Cesarean Section (CS) is a common obstetric surgery that can be performed by both general or regional anaesthetic techniques. Hypotension is the most common complication of spinal anaesthesia, its incidence varying from 70% to 80 %, if severe, it can result in serious perinatal adverse outcomes, such as maternal nausea and vomiting, fetal acidosis and may be an important contributory factor for maternal death related to regional anaesthesia.

DETAILED DESCRIPTION:
A variety of methods have been used for the prevention of post-spinal hypotension which includes the use of intravenous fluid, vasopressors, and physical methods such as table tilt, leg binders, and compression devices. However, a single technique is ineffective and a combination of interventions is suggested.

A care bundle is a group of three to five evidence-based interventions that, when performed together, have a better outcome than if performed individually. A care bundle consists of a group of (usually) between three and five evidence-based interventions. These are related to a particular condition or event for patient care.

Care bundles are well known in the field of intensive care medicine such as Ventilator-Associated Pneumonia (VAP) care bundle, sepsis care bundle, and Central Line-Associated Bloodstream Infection (CLABSI) care bundle.

To our knowledge, till now, no one has investigated a special care bundle in the field of anaesthesia.

In this work, we will investigate the safety and efficacy of a special care bundle in controlling spinal induced hypotension.

ELIGIBILITY:
Inclusion Criteria:

* Age more than 21 years old and less than 40 years.
* Patients are ASA I (American Society of Anesthesiology physical status Grade I) = (normal healthy patients) or ASA II (American Society of Anesthesiologists physical status Grade II) = (patients with mild systemic disease and no functional limitations).
* None laboring, at term with singleton uncomplicated pregnancies.
* Delivery under spinal anesthesia, with height 150 to 180 cm
* Body mass index of at most 40 kg/m2.

Exclusion Criteria:

* Parturient with peri-partum disorders as DM, HTN, cardiac diseases, bronchial asthma or bleeding disorders
* Obesity: BMI >40
* Any known allergy to local anesthetic drugs or ondansetron.
* Apparent anatomical abnormalities or infections in the back region.
* Bleeding disorders e.g., thrombocytopenia, high INR, high PT in the chronic liver or impaired kidney).
* Refusal to participate in the study

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-11-20 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
consumption of ephedrine | immediately at the end of the surgery
  The total consumption of ephedrine used to manage the spinal induced hypotension with CS

SECONDARY OUTCOMES:
consumption of atropine | immediately at the end of the surgery
  The total consumption of atropine used to manage the spinal induced hypotension with CS
postspinal hypotension | immediately at the end of the surgery
  The incidence of postspinal hypotension in CS

CONTACTS AND LOCATIONS:
Overall Officials: Abdelrhman Alshawadfy, Principal Investigator — Suez Canal University
Locations (1):
- Suez Canal University, Ismailia, Egypt